CLINICAL TRIAL: NCT06916169
Title: An Open-label, Randomized, Fasting, Single, Group 2, Stage 2, Cross-over Study to Evaluate the Safety and Pharmacokinetics of AG2304 Compared to Coadministration of AG23041 and AG23042 in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of AG2304 Compared to Coadministration of AG23041 and AG23042
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AG2304 BE
Record Dates: First submitted 2025-04-02; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: Coadministration of AG23041 and AG23042, Period 2: AG2304
  Interventions: Drug: AG2304; Drug: AG23041 and AG23042
- Sequence B (Active Comparator): Period 1: AG2304, Period 2: Coadministration of AG23041 and AG23042
  Interventions: Drug: AG2304; Drug: AG23041 and AG23042

INTERVENTIONS:
Drug: AG2304 — AG2304, Single-dose Oral Administration
Drug: AG23041 and AG23042 — AG23041/AG23042, Single-dose Oral Administration

SUMMARY:
The objective of this study is to evaluate the pharmacokinetic characteristics of AG2304 in healthy subjects.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetic characteristics and safety profiles of AG2304 compared with coadministration AG23041 and AG23042 after a single oral dose administration in healthy Korean subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* A healthy adults aged 19-65 years at the time of screening
* Subjects who are deemed eligible based on the screening tests

Exclusion Criteria:

* Subjects who have taken the investigational drug within 6 months prior to the first dose
* Other exclusions have been applied

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
AUC | Pharmacokinetic plasma samples collected over a 72-hour period
  Area under the plasma concentration
Cmax | Pharmacokinetic plasma samples collected over a 72-hour period
  Peak Plasma Concentration